CLINICAL TRIAL: NCT01002742
Title: A Multi-Center, Randomized, Double Blind, Phase III Trial Evaluating Corticosteroids With Mycophenolate Mofetil vs. Corticosteroids With Placebo as Initial Systemic Treatment of Acute Graft-Vs-Host-Disease (BMT CTN #0802)
Brief Title: Acute Graft-versus-Host Disease Treatment (BMT CTN 0802)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMTCTN0802; U01HL069294 (NIH); BMT CTN 0802 (Other: Blood and Marrow Transplant Clinical Trials Network); U01HL069294-06 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Graft-versus-Host Disease; Immune System Disorders
Keywords: GVHD
MeSH Terms: conditions — Graft vs Host Disease; Immune System Diseases | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Experimental): Corticosteroids with placebo
  Interventions: Drug: Placebo
- Mycophenolate Mofetil (Experimental): Corticosteroids with Mycophenolate Mofetil
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Oral dosing should be delivered in 250 mg units. For those < 40 kg, IV dosing should be within ± 10% of the exact dose. Intravenous doses are infused over a two-hour period.
  * Patients who weight > 60 kg should receive MMF 1 gm PO/IV every 8 hours.
  * Patients who weight between 40-60 kg should receive 750 mg PO/IV every 8 hours.
  * Patients who weight <40 kg should receive 20 mg/kg IV or PO every 8 hours.
  Other Names: Cellcept®; MMF
  Arms: Mycophenolate Mofetil
Drug: Placebo — Oral dosing should be delivered in 250 mg units blinded placebo. For those < 40 kg, IV dosing should be within ± 10% of the exact dose. Intravenous doses are infused over a two-hour period.
  * Patients who weight > 60 kg should receive placebo 1 gm PO/IV every 8 hours.
  * Patients who weight between 40-60 kg should receive 750 mg PO/IV every 8 hours.
  * Patients who weight <40 kg should receive 20 mg/kg IV or PO every 8 hours.
  Other Names: Inactive drug
  Arms: Placebo

SUMMARY:
The study is a Phase III, randomized double blind, placebo controlled, and trial evaluating the addition of Mycophenolate mofetil (MMF) vs. placebo to systemic corticosteroids as initial therapy for acute Graft Vs Host Disease (GVHD). The primary endpoint will be GVHD free survival at Day 56 post randomization.

DETAILED DESCRIPTION:
Corticosteroids have been used as primary therapy for acute GVHD for many years. Historical published and unpublished data from Johns Hopkins, M. D. Anderson, University of Michigan and others defined an expected 35%-53% complete response (CR) at Day +28 of corticosteroid therapy for previously untreated patients with acute GVHD.

BMT CTN study 0302 (NCT00224874)was a randomized Phase II study evaluating etanercept, mycophenolate mofetil, denileukin diftitox or pentostatin in addition to corticosteroids. The results of that study suggested that mycophenolate mofetil produced the highest rates of CR at Day 28 and overall survival, supporting its evaluation in a Phase III study. Day 56 GVHD-free survival for the four treatment arms (all combining corticosteroids with one of the four study drugs) ranged from 39-71% across the four study arms.

ELIGIBILITY:
Inclusion Criteria:

* Acute GVHD developing after allogeneic hematopoietic stem cell transplant using either bone marrow, peripheral blood stem cells or cord blood. Recipients of non-myeloablative and myeloablative transplants are eligible.
* Acute GVHD after planned donor lymphocyte infusion or planned T cell add back are eligible.
* De novo acute GVHD requiring systemic therapy. GVHD is defined as the presence of skin rash and/or persistent nausea, vomiting, and/or diarrhea and/or cholestasis presenting in a context in which acute GVHD is likely to occur and where other etiologies such as drug rash, enteric infection, or hepatotoxic syndromes are unlikely or have been ruled out. Note that patients with stage I and II skin only (overall grade I) or isolated upper gastrointestinal (GI) involvement are eligible if the treating physician deems that systemic high-dose corticosteroid treatment is indicated.
* The patient must have had no previous systemic immune suppressive therapy for treatment of acute GVHD except for a maximum 72 hours of prior corticosteroid therapy at >0.5mg/kg methylprednisolone or equivalent after the onset of acute GVHD.
* Clinical status at enrollment to allow tapering of steroids to not less than 0.25 mg/kg/day prednisone (0.2 mg/kg/day methylprednisolone) at Day 28 of therapy.
* Absolute neutrophil count (ANC) greater than 500/µL.
* Written informed consent and/or assent from patient, parent or guardian.
* Documentation that the assent document and education materials have been provided to, and reviewed with, patients between the ages of 7 and 17.
* Patients of all ages are eligible.
* Biopsy confirmation of GVHD is recommended, but not required. Enrollment should not be delayed for biopsy or pathology results unless these are to be used to decide about whether to treat for GVHD.

Exclusion Criteria:

* Patients receiving mycophenolate mofetil or mycophenolic acid (Myfortic) within seven days of screening for enrollment.
* Patients with uncontrolled infections will be excluded. If a bacterial or viral infection is present, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. If a fungal infection is present, patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Relapsed/persistent malignancy requiring rapid immune suppression withdrawal.
* Patients with GVHD after an unplanned Donor Lymphocyte Infusion (DLI), i.e., DLI that was not part of their original transplant therapy plan, or DLI given for treatment of persistent or recurrent malignancy after transplantation.
* Patients unlikely to be available at the transplantation center on Day 28 and 56 of therapy.
* A clinical syndrome resembling de novo chronic GVHD developing at any time after allotransplantation.
* Patients receiving other drugs for the treatment of GVHD.
* Patients receiving methylprednisolone > 0.5 mg/kg/day (or 0.6 mg/kg/day prednisone) within 7 days before the onset of acute GVHD. If steroid therapy has been administered for treatment of a non-GVHD related condition and tapered to ≤ 0.5 mg/kg/day methylprednisolone (0.6 mg/kg/day prednisone) for seven or more days before the onset of acute GVHD, the patient is eligible.
* Patients who are pregnant, breast feeding, or, if sexually active, unwilling to use effective birth control for the duration of the study. Available evidence and/or expert consensus is inconclusive or is inadequate for determining infant risk when used during breastfeeding, therefore breast feeding patients are not eligible.
* Adults unable to provide informed consent.
* Patients on dialysis.
* Patients with severe hepatic Veno-Occlusive Disease (VOD) or sinusoidal obstruction syndrome who in the judgement of the treating physician are not expected to have normalized bilirubin by Day 56 after enrollment.
* Patients with a history of intolerance/allergy to MMF.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (36):
- United States (36):
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego Medical Center, La Jolla, California
  - Stanford Hospital and Clinics, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Florida College of Medicine, Gainesville, Florida
  - BMT Program at Northside Hospital, Atlanta, Georgia
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Indiana BMT at Beech Grove, Beech Grove, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Maryland Medical Systems, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - DFCI, Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, Barnes Jewish Hospital, St Louis, Missouri
  - Hackensack Univ. Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, NY Presbyterian Hospital, New York, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Levine Children's Hospital, Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Hematology & Transplant Center, Sioux Falls, South Dakota
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas, MD Anderson Cancer Research Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Findings will be published in a manuscript.
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Bolanos-Meade J, Logan BR, Alousi AM, Antin JH, Barowski K, Carter SL, Goldstein SC, Hexner EO, Horowitz MM, Lee SJ, Levine JE, MacMillan ML, Martin PJ, Mendizabal AM, Nakamura R, Pasquini MC, Weisdorf DJ, Westervelt P, Ho VT. Phase 3 clinical trial of steroids/mycophenolate mofetil vs steroids/placebo as therapy for acute GVHD: BMT CTN 0802. Blood. 2014 Nov 20;124(22):3221-7; quiz 3335. doi: 10.1182/blood-2014-06-577023. Epub 2014 Aug 28. PMID 25170121
- [Derived] Shah O, Tamaresis JS, Kenyon LJ, Xu L, Zheng P, Gupta P, Rangarajan K, Lee S, Spellman S, Nikiforow S, Zehnder J, Meyer EH. Analysis of the Whole CDR3 T Cell Receptor Repertoire after Hematopoietic Stem Cell Transplantation in 2 Clinical Cohorts. Biol Blood Marrow Transplant. 2020 Jun;26(6):1050-1070. doi: 10.1016/j.bbmt.2020.01.020. Epub 2020 Feb 18. PMID 32081787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from February 17, 2010 to November 11, 2011 from 36 different transplant centers.
Period: Overall Study
Arm/Group | Placebo | Mycophenolate Mofetil
Started | 119 | 117
Completed | 119 | 116
Not Completed | 0 | 1
Not completed — Determined to be ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients were included in primary, intention-to-treat analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mycophenolate Mofetil | Total
Number analyzed (Participants) | 119 | 116 | 235
Age, Customized [Median (Full Range); unit: years]
  Median Age | 52.9 [9.1 to 76.3] | 54 [9.1 to 76.36] | 53.8 [9.1 to 76.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 45 | 86
  Male | 78 | 71 | 149
Primary Disease [Number; unit: participants]
  Acute myeloid leukemia | 47 | 41 | 88
  Acute lymphoblastic leukemia | 14 | 16 | 30
  Chronic myeloid leukemia | 5 | 3 | 8
  Myelodysplastic syndrome | 17 | 20 | 37
  Lymphoma | 17 | 17 | 34
  Other | 19 | 19 | 38
Unrelated Donor [Number; unit: participants] — Not all participants were matched with an unrelated donor.
  participants | 72 | 66 | 138
Graft Source [Number; unit: participants]
  Bone marrow | 16 | 23 | 39
  Peripheral blood stem cell | 102 | 91 | 193
  Cord blood | 1 | 2 | 3
Myeloablative Conditioning [Number; unit: participants] — Not all participants received Myeloablative Conditioning.
  participants | 74 | 74 | 148
Grade of acute Graft-Vs-Host-Disease (GVHD) at Diagnosis [Number; unit: participants] — Participants are graded on a scale of 1 to 4 according to their symptoms and organs involved, where 4 represents a worse grade.
  participants
    Grade I | 16 | 11 | 27
    Grade II | 62 | 68 | 130
    Grade III | 34 | 30 | 64
    Grade IV | 7 | 7 | 14
Cutaneous involvement at onset [Number; unit: participants]
  No Rash | 36 | 31 | 67
  Maculopapular Rash, <25% of Body Surface | 14 | 11 | 25
  Maculopapular Rash, 25-50% of Body Surface | 21 | 27 | 48
  Generalized Erythroderma | 44 | 46 | 90
  Erythroderma and Bullae Formation/Desquamation | 4 | 1 | 5
Upper GI Abnormalities at Diagnosis [Number; unit: participants]
  No Protracted Nausea and Vomiting | 82 | 85 | 167
  Persistent Nausea, Vomiting or Anorexia | 37 | 31 | 68
Lower GI Abnormalities at Diagnosis [Number; unit: participants]
  No Diarrhea | 66 | 57 | 123
  Diarrhea Less ≤ 500 mL/day | 19 | 21 | 40
  Diarrhea >500 but ≤ 1000 mL/day | 14 | 21 | 35
  Diarrhea >1000 but ≤ 1500 mL/day | 9 | 8 | 17
  Diarrhea >1500 mL/day | 11 | 7 | 18
  Stool with Frank Blood or Melena | 0 | 2 | 2
Liver Abnormalities at Diagnosis [Number; unit: participants]
  Bilirubin <2 mg/dL | 110 | 106 | 216
  Bilirubin 2-3 mg/dL | 5 | 1 | 6
  Bilirubin 3.1-6 mg/dL | 4 | 6 | 10
  Bilirubin 6.1-15 mg/dL | 0 | 2 | 2
  Bilirubin >15 mg/dL | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: GVHD-free Survival
Description: Success is defined as alive and free of GVHD at day 56 after randomization, all others are considered to be a study failure.
Time Frame: Day 56
Measure: Number; unit: participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
participants
  GVHD free | 60 | 69
  Study Failure | 59 | 47

2. Secondary Outcome: Percentage of Surviving Participants With Complete Response (CR)
Description: CR is defined as a score of 0 for the GVHD grading in all evaluable organs.
Time Frame: Days 14, 28, and 56
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
percentage of participants
  Day 14 | 49.6 | 44
  Day 28 | 44.5 | 46.6
  Day 56 | 53.8 | 60.3

3. Secondary Outcome: Incidence of GVHD Flares Requiring Increased Therapy
Description: Flares are defined as any progression of acute GVHD after an initial response (i.e., earlier CR or PR) that requires re-escalation of steroid dosing, or initiation of additional topical or systemic therapy.
Time Frame: Day 90
Measure: Number; unit: participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
participants | 16 | 8

4. Secondary Outcome: Incidence of Discontinuation of Immune Suppression Without Flare
Time Frame: Day 56, Day 180 and Day 360 post-treatment
Population: No data collected
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cumulative Steroid Dose
Description: The cumulative steroid dose for each patient will be calculated by adding the doses (end of each week's dose) for each of the first four weeks of treatment, divided by the number of days of survival during this interval. The cumulative steroid dose was calculated for all patients per treatment arm and compared.
Time Frame: Days 28 and 56
Measure: Number; unit: mg/kg
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
mg/kg
  Day 28 | 0.63 | 0.60
  Day 56 | 0.20 | 0.17

6. Secondary Outcome: Incidence of Topical/Non-absorbable Therapy
Time Frame: Day 56
Measure: Number; unit: participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
participants | 81 | 77

7. Secondary Outcome: Overall GVHD-free Survival Post-randomization
Time Frame: Months 6 and 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
percentage of participants
  6 Months | 73.4 [64.4 to 80.5] | 72.0 [62.8 to 79.3]
  12 Months | 64.7 [55.2 to 72.6] | 57.8 [48.2 to 66.3]

8. Secondary Outcome: Incidence of Chronic GVHD
Time Frame: 12 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
percentage of participants | 43.3 [34.2 to 52.4] | 41.5 [32.3 to 50.7]

9. Secondary Outcome: Incidence of Systemic Infections
Description: Number of participants that experienced at least one infection.
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
participants | 77 | 81

10. Secondary Outcome: Incidence of Epstein-Barr Virus (EBV)-Associated Lymphoma
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
participants | 4 | 6

11. Secondary Outcome: Incidence of Cytomegalovirus (CMV) Reactivation
Time Frame: Year 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
percentage of participants | 39 | 44

12. Secondary Outcome: Cumulative Incidence of a Severe/Life-threatening/Fatal Infections
Time Frame: Year 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
percentage of participants | 42.9 [33.9 to 52.0] | 44.5 [35.3 to 53.6]

13. Secondary Outcome: Disease-Free Survival (DFS) Post-Randomization
Description: DFS includes death or progression/relapse of malignancy
Time Frame: Year 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
percentage of participants | 63 [53.6 to 71.1] | 53.9 [44.4 to 62.5]

14. Secondary Outcome: Treatment Related Mortality (TRM)
Time Frame: Year 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 119 | 116
percentage of participants | 21.5 [14.0 to 29.0] | 21.8 [14.2 to 29.4]

15. Secondary Outcome: Change in Patient Reported Outcomes From Enrollment to Day 56
Time Frame: Day 56
Population: No data collected
Arm/Group | Placebo | Mycophenolate Mofetil
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year following initiation of therapy.
Description: Serious adverse events are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event.
Arm/Group | Placebo | Mycophenolate Mofetil
Serious Adverse Events (participants affected / at risk) | 13/119 | 13/116
Other Adverse Events (participants affected / at risk) | 0/119 | 0/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=119) | Mycophenolate Mofetil (N=116)
Vomiting (Gastrointestinal disorders) | 0 | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 (1)
Cerebellar ataxia (Nervous system disorders) | 0 | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Syncope (Nervous system disorders) | 0 | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Renal failure (Renal and urinary disorders) | 0 | 1 (1)
Sepsis (Infections and infestations) | 0 | 1 (1)
Transaminases increased (Investigations) | 0 | 1 (1)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1) | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0
Septic shock (Infections and infestations) | 2 (2) | 0
Haematuria (Renal and urinary disorders) | 3 (3) | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0
Vertebroplasty (Surgical and medical procedures) | 1 (1) | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-01-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT01002742/Prot_SAP_ICF_000.pdf